CLINICAL TRIAL: NCT05461846
Title: Effect of Integrated Neuromuscular Inhibition Technique on Pain, Function and Muscle Activity in Females With Menstrual Low Back Pain
Brief Title: Effect of Integrated Neuromuscular Inhibition Technique in Females With Menstrual Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Hamdy, lecturer of pt for basic science, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p.T.RCE/012/003493
Record Dates: First submitted 2022-07-11; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): The integrated neuromuscular inhibition technique (INIT) is a manual deactivation trigger points technique and includes the application of ischemic pressure and stretch, the muscle energy technique and the Strain-counterstrain technique.
  Interventions: Other: integrated neuromuscular inhibition technique
- Group (B) (No Intervention): control group

INTERVENTIONS:
Other: integrated neuromuscular inhibition technique — is a manual deactivation trigger points technique and includes the application of ischemic pressure and stretch, the muscle energy technique and the Strain-counterstrain technique.
  Arms: Group (A)

SUMMARY:
Dysmenorrhea is a common problem in women of reproductive age. Primary dysmenorrhea is defined as recurrent, cramping pain occurring with menses in the absence of identifiable pelvic pathology .

DETAILED DESCRIPTION:
Primary dysmenorrhea is characterized by a crampy supra-pubic pain that begins somewhere between several hours before and a few hours after the onset of the menstrual bleeding. Symptoms peak with maximum blood flow and usually last less than one day, but the pain may persist up to 2 to 3 days. Symptoms are more or less reproducible from one menstrual period to the other. The pain is characteristically colicky and located in the midline of the lower abdomen and may extend to lower quadrants, the lumbar area, and the thighs.

Menstrual low back pain (LBP) is one of the common complaints among women. Previous studies have indicated that more than 40% to 50% of the population experience LBP during the menstrual phase (days 1-6) of the menstrual cycle .

ELIGIBILITY:
Inclusion Criteria:

1. Thirty adolescent females suffering from menstrual low back pain.
2. Their age will be ranged from 17 to 24 years.
3. Their body mass index will be ranged from 20 to 25 kg/m2.

Exclusion Criteria:

1. Personal and individual differences between the subjects.
2. Psychological and physical status of subjects which may affect the treatment and evaluation stage.
3. Environmental factors which may affect the subject's response

Ages: 17 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | up to 2 months
  The pain intensity will be assessed through visual analogue scale (VAS) for both groups before and after the end of treatment program. Each woman will be asked to mark a point on the line between the extremes that related to her pain intensity.

SECONDARY OUTCOMES:
function | up to 2 months
  Oswestery Disability Index will be used to assess level of functional disability for both groups before and at the end of the study
muscle amplitude in the form of normalized root mean square (RMS) | up to 2 months
  muscle amplitude will be measured by surface electromyography for upper trapezius

IPD SHARING:
Plan to Share IPD: Undecided